CLINICAL TRIAL: NCT02224014
Title: Lendormin D® Tablet (Drug Use Result Survey)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 263.509
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Sleep Initiation and Maintenance Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Lendormin D tablets
  Interventions: Drug: Lendormin D tablets

INTERVENTIONS:
Drug: Lendormin D tablets

SUMMARY:
Study to investigate the safety and the efficacy in patients with insomnia, receiving Lendormin D tablet under condition of normal clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with insomnia

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with insomnia, receiving Lendormin D tablet under condition of normal clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 485 (Actual)
Dates: Start 2005-06; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to 2 months
Number of patients with adverse drug reactions | up to 2 months
Number of patients with serious adverse events | up to 2 months

SECONDARY OUTCOMES:
Physician's overall efficacy assessment on a 3-point scale | up to 2 months
Patient's impression questionnaire | up to 2 months